CLINICAL TRIAL: NCT04218812
Title: Prospective Multicenter Study on Localization Accuracy and Clinical Utility of Automated Electric Source Imaging in Presurgical Evaluation( PROMAESIS)
Brief Title: Clinical Utility of Automated Electric Source Imaging in Presurgical Evaluation
Acronym: PROMAESIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sándor Beniczky (Other)
Collaborators: Filadelfia Epilepsy Hospital (Other); Hospital del Mar (Other); Brno Epilepsy Center (Unknown); University Hospital Bucharest (Adult) (Unknown); Freiburg University (Unknown); Kepler University Clinic, Linz (Unknown); Motol University Hospital (Other); Christian Doppler Klinik, Salzburg (Unknown); Unidade Local de Saúde de Coimbra, EPE (Other); Valencia University Hospital (Unknown); Carlo Besta Institure, Milano (Unknown); Hospital de Santa Maria, Lisbon (Unknown)
Responsible Party: Sponsor-Investigator, Sándor Beniczky, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PROMAESIS
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Electroencephalography; Refractory Epilepsy; Brain Imaging; Surgery
Keywords: Sensitivity; Specificity; Accuracy; Automated ESI; Refractory epilepsy; Epilepsy surgery; Clinical Utility
MeSH Terms: conditions — Drug Resistant Epilepsy; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Evaluation of automated electrical source imaging(ESI) in epilepsy surgery.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No electrical source imaging (ESI) (Active Comparator): The multidisciplinary teams take decisions based on considering all data without ESI
  Interventions: Diagnostic Test: No electrical source imaging (ESI); Diagnostic Test: Automated electrical source imaging (ESI)
- Automated Electrical source imaging (ESI) (Experimental): The multidisciplinary teams take decisions based on considering all data with ESI
  Interventions: Diagnostic Test: No electrical source imaging (ESI); Diagnostic Test: Automated electrical source imaging (ESI)

INTERVENTIONS:
Diagnostic Test: No electrical source imaging (ESI) — For all patients: MRI, semiology, visual interpretation of EEG, and in selected cases, PET, SPECT
Diagnostic Test: Automated electrical source imaging (ESI) — The automated source imaging consists of 2 phases
  1. Automated detection of EDs
  2. Source imaging of each spike cluster and seizure onset epoch.

SUMMARY:
Electrical source imaging is part of the presurgical evaluation of patients with drug-resistant focal epilepsy. The software packages that will be used in this study have Declaration of Conformity within the European Economic Area (CE mark) for this specific medical use. In spite of being part of the clinical standard, the evidence for the accuracy and clinical utility of these methods are derived from several smaller-scale and retrospective studies. The PROMAESIS study will provide solid evidence of the accuracy and clinical utility of automated ESI.

DETAILED DESCRIPTION:
One-third of patients with epilepsy have seizures resistant to pharmacotherapy. There are many approaches developed to control these seizures, yet epilepsy surgery is still the most common method. The crucial part of epilepsy surgery is to assess the epileptic zone in order to render patients seizure free. However, accurate localization of the epileptic zone is often challenging due to the multimodal approach. This contains semiology, EEG (obtained during long term video-EEG monitoring), magnetic resonance Imaging (MRI), in addition to certain cases, positron emission computed tomography (PET), and single photon emission computed tomography (SPECT) and magnetoencephalography (MEG). At present, in one of the third patients, seizure remains after epilepsy surgery. Therefore a new preoperative method should be improved to assess the epileptic zone. Automated ESI is a post-processing novel method that estimates the location in the brain of the source of the recorded EEG signals.

The objective of this study is:

1. To determine the accuracy of ESI in localizing the epileptic focus.
2. To determine the clinical utility of ESI on clinical decision making

Methods:

Study design: a prospective diagnostic study in line with the Standards for Reporting Diagnostic Accuracy Studies (STARD).

EEG was recorded using the International Federation of Clinical Neurophysiology (IFCN) electrode array of 25 electrodes including six electrodes in the Inferior temporal chain (F9/10, T9/10, and P9/10) in addition to the 19 electrodes of the 10-20 system. Electrode impedance was kept below 5 kilo-ohm. EEG was recorded with a sampling frequency of 256 Hz. The investigators will make a video on how to place the electrodes, to make sure all centers follow a standardized method. Multidisciplinary epilepsy teams classify that in the first step you should keep the multidisciplinary team blinded to the source imaging data, and make the implantation plan without the ESI results. Then show the ESI, adjust the plan and note the changes.

The multidisciplinary teams in different centers will classify seizures into "types." A seizure type is a group of seizures that have stereotypical semiology and ictal EEG. Maximum 3 seizures are registered for per type. After Long Term Monitoring, they provide Epilog and Brain Electrical Source Analysis (BESA) teams with datasets including MRI and Long Term Monitoring recording for each patient. For uploading datasets, multicenter teams will use the platform developed by Epilog. Afterward, Epilog and BESA teams (blinded to patient information) will run the automated source imaging-both for interictal epileptiform discharge (EDs) and ictal signs. Both software packages have CE mark for ESI. Finally, the multidisciplinary teams take decisions in two steps:

I. Considering all data, except ESI II. Adding ESI to all other data.

At each step, the decisions are classified into one of the following categories:

1. Stop (operation not recommended)
2. Implantation of intracranial electrodes
3. Operation

In addition, the changes are classified into one of the following categories:

1. No change - but concordant with the decision.
2. No change - but discordant with decision.
3. Change from stop to implantation.
4. Change from implantation to stop.
5. Change in implantation plan: implantation of additional sites (besides the ones planned in step-1).
6. Change from implantation of operation.
7. Change from operation to implantation.
8. Other (specify in free text). If changes are not related to all analyses results, it will be noted, which method(s) triggered the change (SLORETA-interictal / ictal; Equivalent Current Dipole - interictal/ictal; CLARA interictal/ictal).

At one-year follow-up, the changes are categorized as useful or not useful. A change is defined useful as follows: (a) change from stop to Intracranial Recording: the Intracranial Recording localized the source; (b) change in implantation strategy: the electrode(s) implanted based on the source imaging identified the source; (c) change from implantation to operation: the patient became seizure-free.

ELIGIBILITY:
Inclusion Criteria:

* Patients with drug resistant focal epilepsy, admitted to Epilepsy Monitoring Unit for presurgical evaluation, who are afterwards discussed at the multidisciplinary epilepsy surgery team meetings.

Exclusion Criteria:

* Patients who did not have a seizure during the monitoring.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The Sensitivity and Specificity of automated ESI in presurgical evaluation. | 2 Years
  For determining the the accuracy (sensitivity and specificity) of automated ESI, one year outcome after the operation will be calculated based on the defined criteria.
  * True Positive (TP): source is in the same sub-lobar region as the resection, seizure-free outcome
  * False Positive (FP): source is in the same sub-lobar region as the resection, not seizure-free outcome
  * True Negative (TN): source outside the sub-lobar region that was resected, not seizure-free outcome
  * False Negative (FN): source outside the sub-lobar region that was resected, seizure-free outcome.
the clinical utility of ESI in management of the patient with medically refractory epilepsy | 2 years
  For determining the clinical utility, the percentage of patients in whom automated ESI change decision on patients management will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Rocamora, MD, Principal Investigator — Hospital del Mar; Martin Pali, MD, Principal Investigator — Brno Epilepsy Center; Ioana Mindruta, MD, Principal Investigator — University Hospital Bucharest (Adult); Andreas Schulze Bonhage, MD, Principal Investigator — Freiburg University; Tim von Oertzen, MD, Principal Investigator — Kepler University Clinic, Linz; Vdym Gnatkovsky, MD, Principal Investigator — Carlo Besta Institure, Milano; Peter Marusic, MD, Principal Investigator — Motol University Hospital; Markus Leitinger, MD, Principal Investigator — Christian Doppler Klinik, Salzburg; Francisco Sales, MD, Principal Investigator — Unidade Local de Saúde de Coimbra, EPE; vicente villanueva, MD, Principal Investigator — Valencia University Hospital; Carla Bente, MD, Principal Investigator — Hospital de Santa Maria,
Locations (12):
- Austria (2):
  - Kepler University Clinic, Linz
  - Christian Doppler Klinik, Salzburg
- Czechia (2):
  - Motol University Hospital, Prague, Czech Rebuplic
  - Brno Epilepsy Center, Brno, Czech Republic
- Danish Epilepsy Center, Dianalund, Denmark
- Freiburg University, Freiburg im Breisgau, Baden-Wurttemberg, Germany
- Italy (2):
  - Carlo Besta Institure, Milan
  - Valencia University Hospital, Venice
- Portugal (2):
  - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - Hospital de Santa Maria, Lisbon
- University Hospital Bucharest, Bucharest, Romania
- Hospital del Mar, Barcelona, Spain

REFERENCES:
- [Background] Boon P, D'Have M, Vanrumste B, Van Hoey G, Vonck K, Van Walleghem P, Caemaert J, Achten E, De Reuck J. Ictal source localization in presurgical patients with refractory epilepsy. J Clin Neurophysiol. 2002 Oct;19(5):461-8. doi: 10.1097/00004691-200210000-00009. PMID 12477991
- [Background] Brodbeck V, Spinelli L, Lascano AM, Wissmeier M, Vargas MI, Vulliemoz S, Pollo C, Schaller K, Michel CM, Seeck M. Electroencephalographic source imaging: a prospective study of 152 operated epileptic patients. Brain. 2011 Oct;134(Pt 10):2887-97. doi: 10.1093/brain/awr243. PMID 21975586
- [Background] Beniczky S, Lantz G, Rosenzweig I, Akeson P, Pedersen B, Pinborg LH, Ziebell M, Jespersen B, Fuglsang-Frederiksen A. Source localization of rhythmic ictal EEG activity: a study of diagnostic accuracy following STARD criteria. Epilepsia. 2013 Oct;54(10):1743-52. doi: 10.1111/epi.12339. Epub 2013 Aug 14. PMID 23944234
- [Background] Megevand P, Spinelli L, Genetti M, Brodbeck V, Momjian S, Schaller K, Michel CM, Vulliemoz S, Seeck M. Electric source imaging of interictal activity accurately localises the seizure onset zone. J Neurol Neurosurg Psychiatry. 2014 Jan;85(1):38-43. doi: 10.1136/jnnp-2013-305515. Epub 2013 Jul 30. PMID 23899624
- [Background] Rikir E, Koessler L, Gavaret M, Bartolomei F, Colnat-Coulbois S, Vignal JP, Vespignani H, Ramantani G, Maillard LG. Electrical source imaging in cortical malformation-related epilepsy: a prospective EEG-SEEG concordance study. Epilepsia. 2014 Jun;55(6):918-32. doi: 10.1111/epi.12591. Epub 2014 Apr 4. PMID 24702598
- [Background] Lascano AM, Perneger T, Vulliemoz S, Spinelli L, Garibotto V, Korff CM, Vargas MI, Michel CM, Seeck M. Yield of MRI, high-density electric source imaging (HD-ESI), SPECT and PET in epilepsy surgery candidates. Clin Neurophysiol. 2016 Jan;127(1):150-155. doi: 10.1016/j.clinph.2015.03.025. Epub 2015 May 9. PMID 26021550
- [Background] Maliia MD, Meritam P, Scherg M, Fabricius M, Rubboli G, Mindruta I, Beniczky S. Epileptiform discharge propagation: Analyzing spikes from the onset to the peak. Clin Neurophysiol. 2016 Apr;127(4):2127-33. doi: 10.1016/j.clinph.2015.12.021. Epub 2016 Jan 12. PMID 26818882
- [Background] Mouthaan BE, Rados M, Barsi P, Boon P, Carmichael DW, Carrette E, Craiu D, Cross JH, Diehl B, Dimova P, Fabo D, Francione S, Gaskin V, Gil-Nagel A, Grigoreva E, Guekht A, Hirsch E, Hecimovic H, Helmstaedter C, Jung J, Kalviainen R, Kelemen A, Kimiskidis V, Kobulashvili T, Krsek P, Kuchukhidze G, Larsson PG, Leitinger M, Lossius MI, Luzin R, Malmgren K, Mameniskiene R, Marusic P, Metin B, Ozkara C, Pecina H, Quesada CM, Rugg-Gunn F, Rydenhag B, Ryvlin P, Scholly J, Seeck M, Staack AM, Steinhoff BJ, Stepanov V, Tarta-Arsene O, Trinka E, Uzan M, Vogt VL, Vos SB, Vulliemoz S, Huiskamp G, Leijten FS, Van Eijsden P, Braun KP; E-PILEPSY consortium. Current use of imaging and electromagnetic source localization procedures in epilepsy surgery centers across Europe. Epilepsia. 2016 May;57(5):770-6. doi: 10.1111/epi.13347. Epub 2016 Mar 25. PMID 27012361

DOCUMENTS (1):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT04218812/Prot_001.pdf